CLINICAL TRIAL: NCT05188443
Title: Radiological Imaging in Patients Tested for COVID-19
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 20/WA/0184
Record Dates: First submitted 2022-01-05; First posted 2022-01-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19; Coronary Artery Disease; Cardiovascular Diseases
MeSH Terms: conditions — COVID-19; Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Patients tested for COVID-19 with current or previous (last 3 years) radiological imaging

SUMMARY:
It has become apparent that patients with co-morbidities have an increased risk of mortality from coronarvirus disease 2019 (COVID-19). However, the impact of subclinical respiratory and cardiovascular disease on the outcome of patients with COVID-19 is currently unknown. This observational study will assess the impact of incidental cardiovascular calcification on radiological imaging on the outcomes of patients with COVD-19.

DETAILED DESCRIPTION:
It has become apparent that patients with co-morbidities have an increased risk of mortality from coronarvirus disease 2019 (COVID-19). However, the impact of subclinical respiratory and cardiovascular disease on the outcome of patients with COVID-19 is currently unknown.

Subclinical respiratory and cardiovascular disease can be identified on radiological imaging. For example, calcification in blood vessels can identify cardiovascular disease, intra-thoracic and intra-abdominal fat is associated with coronary artery disease, and lung diseases can be identified on CT and x-ray. The impact these radiological features on the outcomes of patients with COVID-19 is currently unknown.

This study aims to assess the radiological imaging of patients tested for COVID-19 in order to identify the presence of co-existing respiratory and cardiovascular disease and assess their impact on clinical outcomes.

All patients tested for COVID-19 with current or previous (last 3 years) radiological imaging will be included in this study. Radiological images will be de-identified and assessed for the presence of cardiovascular calcification. Information on COVID-19 tests and clinical factors will be obtained from routinely collected data. Additional clinical information will be obtained from electronic health records as required.

ELIGIBILITY:
Inclusion Criteria:

* One or more positive RT-PCR test for COVID-19.
* One or more CT or chest x-ray available performed within the last 3 years

Exclusion Criteria:

* No available radiological imaging within the last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Positive RT-PCR test for COVID-19 with radiological imaging available within the last 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 1 month
  All cause mortality

SECONDARY OUTCOMES:
Cardiovascular mortality | 1 month
  Cardiovascular mortality

OTHER OUTCOMES:
Myocardial infarction | 1 month
  Myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not possible due to data collection method.